CLINICAL TRIAL: NCT02478801
Title: Evaluation of Protein Requirements in Male Endurance Athletes
Brief Title: Protein Requirements in Endurance-trained Athlete
Acronym: EP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Moore, Assistant Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IAAO-E
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Increased Metabolic Requirement; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endurance trained (Experimental): subjects will receive different levels of amino acids intakes varying from 0.2 to 2.8 g/kg/day.
  Interventions: Dietary Supplement: amino acids intake

INTERVENTIONS:
Dietary Supplement: amino acids intake — amino acids intakes will be varied at 0.2-2.8 g/kg/day

SUMMARY:
Protein requirements in individuals who participate in endurance-based exercise training have been suggested to be greater than the current recommended dietary allowance (RDA).

Nutritional requirements for dietary amino acids in adults have traditionally been determined utilizing the nitrogen balance technique, which is prone to underestimating protein requirements. As a result, there is a need to re-evaluate recommendations in order to characterize how dietary amino acid needs may be modulated by physical activity.

Recent studies using the minimally invasive indicator amino acid oxidation (IAAO) technique have suggested that protein requirements in young men are at least 50% higher than RDA based on nitrogen balance data.

Therefore, the purpose of this study is to measure the protein requirement in endurance trained adults using the IAAO technique.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male, endurance-trained participants who regularly more than 40 km/week
* Ability to perform the exercise stimulus (20 km run) on metabolic trial.

Exclusion Criteria:

* Inability to meet health and physical activity guidelines according to the physical activity readiness questionnaire (PAR-Q+)
* Inability to adhere to any of the protocol guidelines (i.e. alcohol, caffeine consumption)
* Regular tobacco use
* Illicit drug use

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
13CO2 (carbon dioxide) excretion (μmol/kg/h) | 4 hours / study day

SECONDARY OUTCOMES:
[13C]phenylalanine oxidation (μmol/kg/h) | 4 hours/study day

REFERENCES:
- [Derived] Kato H, Suzuki K, Bannai M, Moore DR. Protein Requirements Are Elevated in Endurance Athletes after Exercise as Determined by the Indicator Amino Acid Oxidation Method. PLoS One. 2016 Jun 20;11(6):e0157406. doi: 10.1371/journal.pone.0157406. eCollection 2016. PMID 27322029